CLINICAL TRIAL: NCT03720444
Title: "Evaluation of the Effectiveness of the MDT Method (Mechanical Diagnosis and Therapy) in the Management of Low Back Pain in the Subacute Phase"
Acronym: Mc-SubLomb
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_ 0269
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Therapeutics; Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDT (mechanical diagnosis and therapy) method
  Interventions: Other: MDT (mechanical diagnosis and therapy) method

INTERVENTIONS:
Other: MDT (mechanical diagnosis and therapy) method — The intervention consists of a first session to carry out an assessment, followed by 4 reassessment sessions

SUMMARY:
The investigators propose to carry out a study evaluating the effectiveness of the MDT method (mechanical diagnosis and therapy) in the subacute phase of common low back pain.

Few studies have specifically evaluated the effectiveness of the MDT method in the subacute phase, a phase that appears to be crucial before the chronicization of low back pain.

The main objective of this study will be to evaluate the pain of patients managed by the MDT method.

The analysis of the main criterion (Visual Analog Scale) will be done using a type individual clinical trial specific: the Single Case Experimental Design or SCED in lines of multiple bases.

This type of study makes it possible to carry out a comparative test on a single subject acting as its own witness in order to obtain an acceptable level of evidence response for that particular patient.

ELIGIBILITY:
Inclusion Criteria:

* Consultant patients at the Picasso physiotherapy practice (5 rue Nina Simone - 44 000 NANTES)
* Aged 18 to 55 years old
* Suffering from common-looking low back pain. Low back pain is defined as pain or localized discomfort under the 12th dorsal vertebrae and above the inner fold buttock, with possible irradiation to the lower limb but not exceeding the knee.
* Evolving for 4 to 12 weeks (subacute period).
* Period preceded by a period of 30 days without low back pain (in order to avoid recurrent low back pain, rather similar to the chronic phase).

Exclusion Criteria:

* Signs of specific low back pain (confirmed or highly suspected diagnosis): fracture, infection, osteoporosis, inflammatory disease, tumor
* Irradiation below the knee
* Patient knowing she is pregnant
* Protected adults
* Patient with proven cognitive impairment
* Patient with a decompensated psychiatric pathology
* Incapacity to consent
* Refusal to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is all patients aged 18 to 55 years who consult with one of the Mc Kenzie physiotherapists participating in the study, for a common low back pain reason between 4 and 12 weeks of evolution.
  The first ten patients consulting one of the physiotherapists involved and meeting the criteria will be recruited. Each patient will receive information about the research and sign a consent.
  Patients with a strong suspicion of specific low back pain will be excluded from the outset.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Evolution over time of patients' pain | 3 months
  The main outcome will be the evolution over time of patients' pain as assessed by a visual analogue scale completed daily by the patient himself.

SECONDARY OUTCOMES:
Evolution of the pain localization will be done on a body chart filled daily by the patient | 3 months
  Evolution of the pain localization will be done on a body chart filled daily by the patient
Evolution of drug consumption through a completed questionnaire daily by the patient | 3 months
  Evolution of drug consumption through a completed questionnaire daily by the patient
Evolution of functional disability through the EIFEL questionnaire | 3 months
  Evolution of functional disability through the EIFEL questionnaire
Evolution of beliefs and fears through the FABQ (Fear Avoidance Belief) questionnaire | 3 months
  Evolution of beliefs and fears through the FABQ (Fear Avoidance Belief) questionnaire
Evolution of psychosocial factors by STarT Back | 3 months
  Evolution of psychosocial factors by STarT Back

CONTACTS AND LOCATIONS:
Overall Officials: Celine BOUTON, Professor, Principal Investigator — Nantes University
Locations (1):
- Picasso physiotherapy cabinet (5 rue Nina Simone - 44 000 NANTES), Nantes, France

IPD SHARING:
Plan to Share IPD: No